CLINICAL TRIAL: NCT04025996
Title: Using the REtina as a Window To Detect Cardiac microvasculAR Dysfunction In Diabetes Mellitus
Brief Title: REWARD: Using the REtina as a Window To Detect Cardiac microvasculAR Dysfunction In Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Singapore National Eye Centre (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017/2592
Record Dates: First submitted 2018-04-04; First posted 2019-07-19 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-09

CONDITIONS: Retinopathy, Diabetic; Diastolic Dysfunction; Microalbuminuria
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diseased Group: Patients with type 2 diabetic retinopathy and known cardiac dysfunction.
  Interventions: Diagnostic Test: Cardiac Assessments and Eye Assessments

INTERVENTIONS:
Diagnostic Test: Cardiac Assessments and Eye Assessments — Cardiac Assessments, include the following:
  * transthoracic echocardiography
  * computed tomography of coronary arteries
  * position emission tomography computed tomography or single photon emission tomography computed tomography
  Eye examinations, include the following:
  * pupil dilation
  * retinal photography
  * dynamic vessel analyser
  * IOL master

SUMMARY:
Retinopathy may be associated with diastolic dysfunction and/or coronary flow reserve in the heart, and albuminuria in diabetic patients. The objective of this study is to examine the cross-sectional relationships of retinopathy with indices of left ventricular diastolic function, coronary flow reserve and urinary albumin excretion, among diabetic patients.

DETAILED DESCRIPTION:
Diabetes is a potent risk factor for macrovascular coronary disease, leading to systolic dysfunction and heart failure. More recently diabetic microvascular disease has been recognized to play a key role in the development of diastolic dysfunction and heart failure with preserved ejection fraction. A new paradigm in diabetic heart disease centers on microvascular endothelial dysfunction involving the intra-myocardial capillaries and leading to cardiomyocyte dysfunction and diastolic dysfunction. This is analogous to the microvascular dysfunction well-described in the diabetic retinopathy and nephropathy. Yet, whereas diabetic retinal screening for retinopathy and screening for microalbuminuria are routine, diabetic cardiac screening for microvascular dysfunction is practically non-existent. The retinal vasculature may represent a window of opportunity to detect concurrent microvascular disease in the heart and kidneys before the onset of clinical symptoms. However, there are limited studies that directly attempt to correlate retinopathy to diastolic dysfunction and microalbuminuria. Hence this study aims to examine the cross-sectional relationships of retinopathy with indices of left ventricular diastolic function, coronary flow reserve and urinary albumin excretion, among diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than equal to 21 years old

Exclusion Criteria:

* Known history of active eye lens or corneal opacity
* Known allergy to eye drops
* Kidney disease with estimated GFR < 60
* Pregnant or lactating women
* Asthmatic status of the moderate persistent and above categories
* Chronic obstructive pulmonary disease
* Thyroid dysfunction

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have known heart condition and type II diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Eye Examination | 1 day
  Retinal photography on diabetic patients will be performed to identify those with retinopathy.
Cross-sectional analyses will be performed to look at the association between diabetic retinopathy with left ventricular diastolic function, coronary flow reserve and urinary albumin excretion. | 2 days
  These data will provide initial evidence of the mechanistic link between microvascular dysfunction in the eye, heart and kidneys among patients with diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phan K, Mitchell P, Liew G, Plant AJ, Wang SB, Au C, Chiha J, Kovoor P, Thiagalingam A, Burlutsky G, Gopinath B. Association between Retinal Arteriolar and Venule Calibre with Prevalent Heart Failure: A Cross-Sectional Study. PLoS One. 2015 Dec 11;10(12):e0144850. doi: 10.1371/journal.pone.0144850. eCollection 2015. PMID 26659133
- [Background] Wong TY, Rosamond W, Chang PP, Couper DJ, Sharrett AR, Hubbard LD, Folsom AR, Klein R. Retinopathy and risk of congestive heart failure. JAMA. 2005 Jan 5;293(1):63-9. doi: 10.1001/jama.293.1.63. PMID 15632337
- [Background] Lam CS, Roger VL, Rodeheffer RJ, Bursi F, Borlaug BA, Ommen SR, Kass DA, Redfield MM. Cardiac structure and ventricular-vascular function in persons with heart failure and preserved ejection fraction from Olmsted County, Minnesota. Circulation. 2007 Apr 17;115(15):1982-90. doi: 10.1161/CIRCULATIONAHA.106.659763. Epub 2007 Apr 2. PMID 17404159
- [Background] Lam CS, Lyass A, Kraigher-Krainer E, Massaro JM, Lee DS, Ho JE, Levy D, Redfield MM, Pieske BM, Benjamin EJ, Vasan RS. Cardiac dysfunction and noncardiac dysfunction as precursors of heart failure with reduced and preserved ejection fraction in the community. Circulation. 2011 Jul 5;124(1):24-30. doi: 10.1161/CIRCULATIONAHA.110.979203. Epub 2011 Jun 13. PMID 21670229
- [Background] Teo LY, Chan LL, Lam CS. Heart failure with preserved ejection fraction in hypertension. Curr Opin Cardiol. 2016 Jul;31(4):410-6. doi: 10.1097/HCO.0000000000000292. PMID 27070649